CLINICAL TRIAL: NCT02735161
Title: Fatigue and Exercise Training in Patients With Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Collaborators: University of Oslo (Other); Hasselt University (Other)
Responsible Party: Principal Investigator, Anne Helene Edvardsen, Head of Out Patient and Laboratory Department, Researcher, LHL Helse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015/23131
Record Dates: First submitted 2016-03-28; First posted 2016-04-12 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Sarcoidosis; Fatigue
Keywords: Sarcoidosis; Fatigue; Exercise
MeSH Terms: conditions — Sarcoidosis; Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise training (Experimental): Four exercise training sessions. Two endurance training sessions, one with high intensity interval training and one session of moderate intensity of longer duration. Two strength training session; one with high load and few repetitions and one with low load and many repetitions.
  Fatigue and lactate will be measured before, after and 24 hours post-exercise. Trainings sessions will be randomized.
  Interventions: Other: Muscle strength training; Other: Endurance exercise training

INTERVENTIONS:
Other: Muscle strength training — Two different muscle strength training protocols will be compared; one exercise session with high load/low repetitions (4 sets x 5RM) versus one exercise session with low load/high repetitions (2 sets x 25RM). Both session will be conducted at four different exercises; seated leg press, chest press, cable lat pull down and seated rowing.
Other: Endurance exercise training — Two different endurance exercise training protocols will be compared; one exercise sessions is interval training with high intensity (85-95% of HRmax) versus one of moderate intensity (70-75% of HRmax) with longer duration.

SUMMARY:
The aims of the current study is to explore if different exercise training protocols affect fatigue post-exercise, and if sarcoidosis-related fatigue and maximal and sub-maximal cardiopulmonary exercise test (CPET) variables change after a 4-weeks exercise training period.

DETAILED DESCRIPTION:
This project aims to provide data on post-exercise fatigue after single exercise sessions with endurance training and muscle strength training, each with two different intensities. For endurance training; post-exercise fatigue will be assessed after one session of high intensity interval training, and one session with longer duration of moderate intensity. For muscle strength training, fatigue will be measured after one session with high loads/few repetitions and one session with low loads/many repetitions. In addition, changes in sub-maximal and maximal metabolic and ventilatory responses to a maximal cardiopulmonary exercise test on a treadmill (CPET) and association to sarcoidosis-related fatigue before and after a 4-weeks exercise training period will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sarcoidosis diagnosed according to the latest American Thoracic Society/European Respiratory Society/World Association for Sarcoidosis and Other Granulomatous Disorders (ATS/ERS/WASOG) statement on sarcoidosis who are attending a four weeks exercise based pulmonary rehabilitation program at LHL-klinikkene Glittre.

Exclusion Criteria:

* Patients with a concurrent and predominant diagnosis of another significant respiratory disorder (for example: asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis, or lung cancer).
* Unstable cardiovascular disease.
* Not able to perform the required physical tests and exercise training sessions caused by co-morbidities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | Fatigue measured immediately before and acute after exercise sessions, (within 1 min.), and addition 24 hours post-exercise.
  Changes of fatigue will be assessed assessed by Visual Analogue Scale (VAS), where the grade of fatigue is assessed between 0 (no fatigue) and 10 (maximal fatigue).

SECONDARY OUTCOMES:
Change in blood lactate | Blood lactate are measured before and acute after exercise sessions (within 2 min.), and in addition 24 hours post-exercise.
  Blood lactate will be assessed by capillary puncture in a finger tip.
Change in sarcoidosis related fatigue | Measured first day and last day of a 4-week exercise based pulmonary rehabilitation
  Assessed by the Fatigue Assessment Scale (FAS)
Change in metabolic and ventilatory variables from CPET | Measured during a CPET first day and last day of a 4-week exercise based pulmonary rehabilitation
  Ratio ventilation/carbon dioxide output (VE/VCO2)
Change in metabolic and ventilatory variables from CPET | Measured during a CPET first day and last day of a 4-week exercise based pulmonary rehabilitation
  Ventilatory (anaerobic) threshold (VT, %)
Change in maximal oxygen uptake | Measured during a CPET first day and last day of a 4-week exercise based pulmonary rehabilitation
  Maximal oxygen uptake (VO2, mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Siri Skumlien, PhD, Study Director — LHL Helse
Locations (1):
- LHL-klinikkene Glittre, Hakadal, Norway

IPD SHARING:
Plan to Share IPD: No